CLINICAL TRIAL: NCT05597579
Title: The Timing of Cognitive Impairments in Psychotic Disorders
Brief Title: Cognitive Impairments in Psychotic Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Mark Weiser, MD, Principal Investigator, Head of Psychiatry, Sheba Medical Center
Other Study IDs: 2974-16-SMC
Record Dates: First submitted 2022-02-24; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Psychotic Disorders; Cognitive Impairment
Keywords: Schizophrenia; Affective Disorders; IQ Tests; Psychotic Disorders; Cognition
MeSH Terms: conditions — Psychotic Disorders; Cognitive Dysfunction; Schizophrenia; Mood Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Patients diagnosed with psychotic disorder.
  Interventions: Diagnostic Test: DAPAR Tests (IQ equivalent test)
- Control Group: Healthy Controls
  Interventions: Diagnostic Test: DAPAR Tests (IQ equivalent test)

INTERVENTIONS:
Diagnostic Test: DAPAR Tests (IQ equivalent test) — This study will compare DAPAR scores before and after the onset of the psychotic illness.

SUMMARY:
Patients with Psychotic disorders (Schizophrenia, Bipolar disorder and Schizoaffective disorder) often suffer from significant cognitive impairments, however how these develop and change over time before and after the first psychotic break is unclear. While there are data by several groups, showing that many future patients have significant cognitive impairments years before the onset of psychosis, many future patients seem to be doing well before the manifestation of psychosis, and decline steeply in functioning after their first psychotic episode. Hence the timing of the onset of cognitive impairment in patients with psychotic disorders requires further exploration. The current study will investigate the timing of cognitive impairment by using IQ tests before and after the first psychotic break

DETAILED DESCRIPTION:
In this study the investigators aim to use the DAPAR tests (A cognitive assessment which all 17 year old Jewish adolescents in Israel undergo to participate in mandatory military service), which measures intelligence, and is equivalent to the IQ test. The subjects will be persons who had their first psychotic break, at least one year following the DAPAR tests. As part of the study, the participants will re-take the DAPAR tests, after the onset of the psychotic illness.

ELIGIBILITY:
Inclusion Criteria - Study Group:

* Patients between the ages 27-18 who had first psychotic break in the last ten years, and more than a year from the date of the DAPAR tests.
* Diagnoses of schizophrenia, Bipolar disorder or Schizoaffective disorder according to DSM-5 criteria.
* Previous DAPAR tests at the age of 17.

Inclusion Criteria - Control group:

* Participants between the ages of 27-18.
* No history of psychotic break.
* Previous DAPAR tests at the age of 17.

Exclusion Criteria - Both groups:

* Participants who did not perform the full battery of the DAPAR tests.
* Participants who have been appointed a guardian.

Exclusion Criteria - Control group:

- Participants who have a first-degree relative who suffers from a psychotic disorder.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The investigators will recruit patients treated in the psychiatric unit at the Sheba Medical Center and in other medical institutions throughout the country. Additionally, subjects will be recruited through internet advertisement of the study. All subjects will give informed consent.
  Control group will be recruited by matching for Age, Sex and socioeconomic status. recruitment will be preforemd by advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in DAPAR (An Israeli cognitive test) scores | 1 day (During recruitment visit)
  Cognitive changes in both groups (lowest 10 - highest 90)

SECONDARY OUTCOMES:
Psychotic Symptoms | 1 day (During recruitment visit)
  PANSS-6 (Positive and Negative Syndrome Scale - Abbrevieted) scores (lowest 0- highest 36)
Social Functioning | 1 day (During recruitment visit)
  PSP (Personal and Social Performance Scale) Scores (lowest 0- highest 100)
Cognitive Functioning | 1 day (During recruitment visit)
  WAIS-III (Wechsler Adult Intelligence Scale) (4 specific sub-tests)
Coping strategies | 1 day (During recruitment visit)
  COPE (Assessing Coping Strategies) scores (lowest 0 - highest 90)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Weiser, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No